CLINICAL TRIAL: NCT01791543
Title: Early Feasibility Study of Intramural Needle Ablation for Ablation of Recurrent Ventricular Tachycardia That Has Failed Conventional Radiofrequency Ablation
Brief Title: Intramural Needle Ablation for Ablation of Recurrent Ventricular Tachycardia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Stevenson (Other)
Responsible Party: Sponsor-Investigator, William Stevenson, Professor, Cardiovascular Medicine, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P000304
Record Dates: First submitted 2013-02-07; First posted 2013-02-15 (Estimated); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Ventricular Tachycardia
Keywords: ventricular tachycardia; ablation; ventricular arrhythmia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intramural Needle Catheter Ablation (Experimental): Ablation of Ventricular Tachycardia with Intramural Needle Ablation Catheter
  Interventions: Device: Intramural Needle Ablation Catheter

INTERVENTIONS:
Device: Intramural Needle Ablation Catheter

SUMMARY:
The purpose of the study is to assess the effectiveness and safety of a new device called an Intramural Needle Ablation Catheter (INA catheter). The INA catheter is used for locating and ablating ventricular arrhythmias that have failed standard radiofrequency ablation. This approach is desirable because some people have ventricular arrhythmias that originate deep within the heart muscle where it is not abolished by ablation with standard catheters.

The investigators seek to determine whether the INA catheter can potentially help people who have ventricular arrhythmias that have failed standard radiofrequency ablation. The investigators also want to determine if it is likely to be safe, without excessive side effects.

ELIGIBILITY:
Inclusion Criteria:

Monomorphic ventricular tachycardia (VT) or incessant ventricular arrhythmia (defined as >20% of beats due to ventricular arrhythmia including unifocal premature ventricular contractions (PVCs ), couplets, nonsustained VT) that is causing a decline in left ventricular (LV) ejection fraction to less than 0.50.

Arrhythmia meets the following criteria:

1. Ventricular arrhythmia is recurrent and symptomatic
2. prior antiarrhythmic drug therapy has failed due to recurrent ventricular arrhythmia, toxicity, or intolerance

   * Age 18 or older
   * Left ventricular (LV) ejection fraction > 0.10 as estimated by echocardiography or contrast ventriculography within the previous 90 days
   * Failed prior VT or PVC ablation due to spontaneous recurrence of the arrhythmia or frequent PVCs.
   * Able and willing to comply with all pre-, post-, and follow-up testing and requirements
   * Signed Informed Consent

Exclusion Criteria:

* Patients with idiopathic VT defined as VT that originates from a region without evidence of scar detected by MRI or voltage mapping in a patient without other evidence of heart disease that is not causing significant depression of ventricular function.
* Definite protruding left ventricular thrombus on pre-ablation echocardiography when LV ablation is required.
* Thrombotic myocardial infarction within the preceding two (2) months.
* Other disease process that is likely to limit survival to less than 12 months.
* Class IV heart failure, unless heart failure is due to frequent or incessant VT.
* Contraindication to heparin.
* Allergy to radiographic contrast dye.
* Severe aortic stenosis
* Severe mitral regurgitation with a flail mitral valve leaflet.
* Significant congenital anomaly or medical problem that in the opinion of the principal investigator would preclude enrollment into the study.
* Enrolled in another investigational study evaluating a drug or device.
* Unstable angina that is not due to frequent or incessant VT.
* Women who are pregnant.
* Thrombocytopenia (platelet count < 50,000) or coagulopathy.
* Acute non-cardiovascular illness or systemic infection.
* Cardiogenic shock unless it is due to incessant VT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Stevenson, M.D., Study Director — Vanderbilt Heart and Vascular Institute; Usha Tedrow, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee

REFERENCES:
- [Background] Sapp JL, Cooper JM, Zei P, Stevenson WG. Large radiofrequency ablation lesions can be created with a retractable infusion-needle catheter. J Cardiovasc Electrophysiol. 2006 Jun;17(6):657-61. doi: 10.1111/j.1540-8167.2006.00439.x. PMID 16836718
- [Background] Sapp JL, Beeckler C, Pike R, Parkash R, Gray CJ, Zeppenfeld K, Kuriachan V, Stevenson WG. Initial human feasibility of infusion needle catheter ablation for refractory ventricular tachycardia. Circulation. 2013 Nov 19;128(21):2289-95. doi: 10.1161/CIRCULATIONAHA.113.003423. Epub 2013 Sep 13. PMID 24036605
- [Background] Schaeffer B, Tanigawa S, Nakamura T, Muthalaly RG, Sapp J, John R, Ghidoli D, Pellegrini C, Tedrow U, Stevenson WG. Characteristics of myocardial tissue staining and lesion creation with an infusion-needle ablation catheter for the treatment of ventricular tachycardia in humans. Heart Rhythm. 2020 Mar;17(3):398-405. doi: 10.1016/j.hrthm.2019.10.007. Epub 2019 Oct 8. PMID 31604127
- [Result] Stevenson WG, Tedrow UB, Reddy V, AbdelWahab A, Dukkipati S, John RM, Fujii A, Schaeffer B, Tanigawa S, Elsokkari I, Koruth J, Nakamura T, Naniwadekar A, Ghidoli D, Pellegrini C, Sapp JL. Infusion Needle Radiofrequency Ablation for Treatment of Refractory Ventricular Arrhythmias. J Am Coll Cardiol. 2019 Apr 2;73(12):1413-1425. doi: 10.1016/j.jacc.2018.12.070. PMID 30922472
- [Derived] Tedrow UB, Kurata M, Kawamura I, Batnyam U, Dukkipati S, Nakamura T, Tanigawa S, Fuji A, Richardson TD, Kanagasundram AN, Koruth JS, John RM, Hasegawa K, Abdelwahab A, Sapp J, Reddy VY, Stevenson WG. Worldwide Experience With an Irrigated Needle Catheter for Ablation of Refractory Ventricular Arrhythmias: Final Report. JACC Clin Electrophysiol. 2023 Aug;9(8 Pt 2):1475-1486. doi: 10.1016/j.jacep.2023.05.014. Epub 2023 May 19. PMID 37278684
- [Derived] Dukkipati SR, Nakamura T, Nakajima I, Oates C, Narui R, Tanigawa S, Sljapic T, Whang W, Koruth JS, Choudry S, Schaeffer B, Fujii A, Tedrow UB, Sapp JL, Stevenson WG, Reddy VY. Intramural Needle Ablation for Refractory Premature Ventricular Contractions. Circ Arrhythm Electrophysiol. 2022 May;15(5):e010020. doi: 10.1161/CIRCEP.121.010020. Epub 2022 Apr 27. PMID 35476455
- [Derived] Qian PC, Oberfeld B, Schaeffer B, Nakamura T, John RM, Sapp JL, Stevenson WG, Tedrow UB. Frequency Content of Unipolar Electrograms May Predict Deep Intramural Excitable Substrate: Insights From Intramural Needle Catheter Ablation of Ventricular Tachycardia. JACC Clin Electrophysiol. 2020 Jul;6(7):760-769. doi: 10.1016/j.jacep.2020.03.003. Epub 2020 Apr 29. PMID 32703556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients referred for ablation of ventricular arrhythmias who met the entry criteria were enrolled at Vanderbilt University Medical Center or Brigham and Women's Hospital from 9/19/2016 to 8/26/2020.
Pre-assignment Details: 115 unique subjects signed consent and were enrolled; 6 were consented twice (121 enrollments): 1 had no needle ablation when standard ablation was successful at both procedures; 3 had needle ablation at the first but not the second procedure; 2 had needle ablation twice and outcomes are reported for their first procedure only. Of the 115, 39 exited before treatment (standard ablation successful in 30, VT not inducible in 7, other reasons in 2). Thus, 76 unique participants started the study.
Groups:
- Intramural Needle Catheter Ablation: Patients meeting the entry criteria and consented for participation in the study
Period: Overall Study
Arm/Group | Intramural Needle Catheter Ablation
Started | 76
Completed | 74
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Intramural Needle Catheter Ablation: Patients Treated With Intramural Needle Ablation
Arm/Group | Intramural Needle Catheter Ablation
Number analyzed (Participants) | 76
Age, Continuous [Median (Full Range); unit: years] | 65 [20 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 76
Left Ventricular Ejection Fraction (LVEF) [Median (Inter-Quartile Range); unit: ejection fraction] — Ejection fraction expressed as a fraction.
  ejection fraction | 0.38 [0.25 to 0.48]
Coronary Artery Disease [Count of Participants; unit: Participants] | 35
Nonischemic heart diseases [Count of Participants; unit: Participants] | 59
History of heart failure [Count of Participants; unit: Participants] | 41
Number of prior failed ablation procedures (median, range) [Median (Full Range); unit: prior procedures] | 2 [1 to 6]
Failed amiodarone [Count of Participants; unit: Participants] | 61
Failed mexiletine [Count of Participants; unit: Participants] | 36
Implanted Defibrillator [Count of Participants; unit: Participants] | 60
Ablation for ventricular tachycardia (VT) [Count of Participants; unit: Participants] | 56
Ablation for premature ventricular contractions (PVCs)/Nonsustained VT [Count of Participants; unit: Participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Without Hospitalization for Ventricular Tachycardia (VT) During 6 Months
Description: Freedom from hospitalization for recurrent Ventricular Tachycardia during the 6 months following ablation for VT.
Time Frame: 6 months
Population: This outcome is analyzed only for the 54 patients whose targeted arrhythmia was ventricular tachycardia.
Measure: Count of Participants; unit: Participants
Groups:
- Intramural Needle Catheter Ablation: Ablation of Ventricular Tachycardia with Intramural Needle Ablation Catheter
  Intramural Needle Ablation Catheter
Arm/Group | Intramural Needle Catheter Ablation
Number analyzed (Participants) | 54
Participants | 38

2. Primary Outcome: Number of Participants With No Serious Adverse Events
Description: Absence of serious adverse events that are potentially device related and occur within 30 days of the ablation procedure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intramural Needle Catheter Ablation
Number analyzed (Participants) | 76
Participants | 63

3. Primary Outcome: Number of Subjects Ablated for Nonsustained Arrhythmias Who Had a Reduction to Less Than 5000 Arrhythmia Beats Daily
Description: Number of subjects who had ablation for nonsustained arrhythmias with ventricular dysfunction who had a decrease in ambient ventricular arrhythmia to < 5000 ventricular beats daily.
Time Frame: 6 months
Population: This outcome is analyzed only for the 20 patients in whom PVCs/Nonsustained VT was the targeted arrhythmia for study entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Intramural Needle Catheter Ablation
Number analyzed (Participants) | 20
Participants | 12

4. Secondary Outcome: Number of Subjects With Acute Abolition of at Least One Clinical Inducible Ventricular Tachycardia or Targeted Nonsustained Arrhythmia
Description: Defined as termination of at least one clinical or presumptive clinical monomorphic VT by Radiofrequency ablation and/or rendering that VT no longer inducible or abolition of a targeted nonsustained arrhythmia.
Time Frame: Baseline to end of the ablation procedure (approximately 5 hours)
Population: This secondary efficacy endpoint was not assessed in 16 patients in whom VT induction was not attempted because in the judgment of the investigator it imposed unwarranted risk of hemodynamic deterioration. Acute success for PVC/nonsustained VT ablation was abolishing the targeted PVC..
Measure: Count of Participants; unit: Participants
Arm/Group | Intramural Needle Catheter Ablation
Number analyzed (Participants) | 60
Participants | 51

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intramural Needle Catheter Ablation
All-Cause Mortality (participants affected / at risk) | 5/76
Serious Adverse Events (participants affected / at risk) | 13/76
Other Adverse Events (participants affected / at risk) | 5/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intramural Needle Catheter Ablation (N=76)
Pericardial Effusion (Cardiac disorders) | 2 (2)
Pulmonary Embolism (Cardiac disorders) | 2 (2)
Retroperitoneal Hematoma (Vascular disorders) | 2 (2)
urinary tract infection (Renal and urinary disorders) | 1 (1)
ventricular fibrillation (Cardiac disorders) | 1 (1) — During catheter manipulation
Allergic reaction (General disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
AV block (Cardiac disorders) | 2 (2)
GI bleed (Gastrointestinal disorders) | 1 (1)
Heart Failure Exacerbation (Cardiac disorders) | 1 (1)
Intraperitoneal bleeding (Gastrointestinal disorders) | 1 (1)
atrial fibrillation with rapid response (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intramural Needle Catheter Ablation (N=76)
Femoral hematoma (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT01791543/Prot_SAP_000.pdf